CLINICAL TRIAL: NCT01714141
Title: Multi-Component Technology Intervention for Minority Emerging Adults With Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Karen MacDonell, PhD, Assistante Professor, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MCTI-1R34HL107664-01A1
Record Dates: First submitted 2012-10-17; First posted 2012-10-25 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Asthma; Poor Medication Adherence
Keywords: Technology based intervention; Emerging adults; African Americans; Asthma; Controller medications; Motivational intervention
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Multi-component, technology based intervention (Experimental): 2 tailored, computer-delivered motivational interviewing sessions targeting adherence to asthma control medications + tailored text messaged reminders to take medications between sessions.
  Interventions: Behavioral: Multi-component, technology based intervention
- Asthma education active control (Active Comparator): Control condition consists of active control matched to intervention for delivery-method and time-- 2 sessions of computer-delivered asthma education + daily text messaged facts about asthma.
  Interventions: Behavioral: Asthma education active control

INTERVENTIONS:
Behavioral: Multi-component, technology based intervention — Motivational sessions were adapted from work done with young adults with HIV (MESA).
  Arms: Multi-component, technology based intervention
Behavioral: Asthma education active control
  Arms: Asthma education active control

SUMMARY:
This pilot study's main goal is to develop and preliminarily test a technology-based intervention to improve asthma medication adherence in urban African American emerging adults (ages 18-29). It is hypothesized that youth randomized to MCTI for adherence will show improvements in motivation to adhere to asthma medications and self-reported adherence compared to the comparison condition at 1- and 3- month follow up.

DETAILED DESCRIPTION:
This study collected pilot data with a sample of 48 African American emerging adults with asthma with suboptimal medication adherence. Half of the sample were randomized to receive a multi-component technology-based intervention (MCTI) targeting adherence to daily controller medication. The MCTI consisted of two components: 1) 2 sessions of computer-delivered motivational interviewing targeting medication adherence, and 2) individualized text messaging focused on medication adherence between the sessions. Text messages were individualized based on Ecological Momentary Assessment (EMA). The remaining half of participants completed a series of computer-delivered asthma education modules matched for length, location, and method of delivery of the intervention session. Control participants also received text messages between intervention sessions. Message content was the same for all control participants and contain general facts about asthma (not tailored).

ELIGIBILITY:
Inclusion Criteria:

African American Live in the Detroit Area, approximately 30 miles from the Hutzel Building Ages 18-29

Have moderate to severe persistent asthma. Persistent asthma is defined according to the 2007 NHLBI guidelines. The level of symptoms, as defined by any of the following in the last 4 weeks:

Use of any asthma medication more than 2 times a week Daytime asthma symptoms such as wheezing, tightness of chest, problems coughing more than 2 times a week, or waking up at night because of asthma more than 2 times a month

Participant is prescribed a daily asthma controller medication, even if they do not take it.

Participant must report poor adherence to daily controller medications during eligibility screening (brief interview).

Poor adherence is defined as not taking medications "as prescribed" less than 4 days per week in any of the 4 weeks prior to enrollment OR as a proxy of poor adherence as self-report of <80% medication adherence in the past 30 days, self-report of emergency room visit/hospitalization for asthma in the past 6 months, or a poor score on the Asthma Control Test.

Participant must be able to complete questionnaires in English Participant must own or have access to a cellular phone for the duration of the study No exclusions will be made due to co-morbid mental health problems (i.e. ADHD, depression) except thought disorders (i.e. schizophrenia, autism), suicidality or mental retardation.

Exclusion Criteria:

Individuals with other chronic health conditions requiring ongoing medical intervention ( e.g., HIV, Type II Diabetes) will be excluded.

These chronic diseases include: Glaucoma, bi-polarism, segmented glomerular nephritis, cystic fibrosis, spondyloarthropathy, congenital heart disease, sickle cell

No pregnant women will be included in this study.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2011-12; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change in medication adherence | baseline, 1 month, 3 month
  Self-reported adherence to asthma controller medication(s) through questionnaire report and, at baseline and 3 months, 7 days of momentary (real time) sampling of adherence behavior via SMS text messaging.
Change in motivation for medication adherence | baseline, 1 month, 3 month
  Self-report of motivation to take asthma controller medications as prescribed.

SECONDARY OUTCOMES:
Change in asthma knowledge | baseline, 1 month, 3 month
  Knowledge of asthma and asthma medications
Change in asthma medication confidence | Baseline, 1 month, 3 month
  Confidence in ability to take asthma medications as prescribed.
Change in asthma medication importance | baseline, 1 month, 3 month
  Perceived importance of taking asthma medication as prescribed.
Change in asthma control | baseline, 1 month, 3 month
  Self-reported asthma control (symptom prevalence, health care utilization)
Change in barriers to taking medication | baseline, 1 month, 3 months
  Self-report of barriers to taking medication. At baseline and 3 months, daily barriers to taking medications as reported in daily diary.
Change in asthma anxiety | baseline, 1 month, 3 month
  Feelings and anxiety associated with living with asthma.
Change in asthma self-efficacy and attitude | baseline, 1 month, 3 month
  Self-report of self-efficacy to manage asthma effectively; attitude towards asthma and asthma management.

REFERENCES:
- [Result] Kolmodin MacDonell K, Naar S, Gibson-Scipio W, Lam P, Secord E. The Detroit Young Adult Asthma Project: Pilot of a Technology-Based Medication Adherence Intervention for African-American Emerging Adults. J Adolesc Health. 2016 Oct;59(4):465-71. doi: 10.1016/j.jadohealth.2016.05.016. Epub 2016 Jul 27. PMID 27475032